CLINICAL TRIAL: NCT05565404
Title: Effect of Mobile Health(mHealth) on Interdental Brushing in Type 2 Embrasures": A Randomized Controlled Clinical Trial.
Brief Title: Effect of mHealth on Interdental Brushing in Type 2 Embrasures"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Jyoti yadav perio 22/26
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis
Keywords: interdental brush; type 2 embrasures; text messages
MeSH Terms: conditions — Periodontitis | interventions — Telemedicine; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Scaling and root planing, interdental brushing demonstration and regular text messages in type 2 embrasure patients.
  Interventions: Behavioral: mobile health
- Control group (Active Comparator): Scaling and root planing, interdental brushing demonstration in type 2 embrasure patients.
  Interventions: Procedure: Scaling and root planing+Interdental aid

INTERVENTIONS:
Behavioral: mobile health — Scaling and root planing, interdental brushing demonstration and regular text messages in type 2 embrasure patients.
  Arms: Test group
Procedure: Scaling and root planing+Interdental aid — Scaling and root planing, interdental brushing demonstration in type 2 embrasure patients.
  Arms: Control group

SUMMARY:
Plaque biofilm is the etiological factor for the development of gingival and periodontal diseases. There are certain areas in mouth where plaque removal is difficult, which includes palatal, lingual and interproximal areas. Among these, interproximal areas are most difficult to clean due to inability of toothbrush to reach that area properly. So, interdental aids are required to remove plaque from the proximal areas efficiently. Consequently, plaque accumulation most often starts in interdental areas, where resultant periodontal lesions are observed most commonly. It is the ethical responsibility of the dental professional to educate patients about the progression of destructive periodontal disease, so that patients understand the need for plaque removal and control. It is not easy for patients to develop any new habits of using different cleaning aids. Many studies have proven mobile health to be effective in improving patient's compliance for better oral hygiene maintenance. So, proper means of education such as mobile health could lead to behavior change and adoption of new habit of using interdental aid on regular basis. Use of mobile technology to track and improve health outcomes is known as mobile health. No studies till date have evaluated mobile health in improving interdental brushing. It is possible that we can reinforce patient on the use of interdental brush with the help of text messages. Therefore, the present randomized controlled clinical trial is designed to evaluate the compliance of interdental brushing with the use of text messages.

DETAILED DESCRIPTION:
Dental plaque is considered to be a biofilm of dynamic and complex microbial community. Microbial composition of plaque varies in every individual and at every site within the same mouth. Plaque accumulation leads to development of gingival and periodontal diseases. It usually takes 7 to 21 days to develop gingivitis in the absence of plaque removal. Plaque control is necessary for maintaining the oral tissues, especially the gingiva, in a healthy state. Primary means of plaque control is through mechanical action, with the toothbrush being the most common means of plaque removal. While it removes plaque efficiently from the buccal, lingual and occlusal surfaces, it fails to do the same at interproximal sites. Consequently, plaque accumulation most often starts in interdental areas, where resultant periodontal lesions are observed most commonly. This makes interdental cleaning very necessary, in addition to toothbrushing, for prevention of gingival and periodontal diseases.

In type 2 embrasure patients, interdental brush is prescribed. It consists of soft nylon filaments twisted into a fine stainless steel wire. These interdental brushes are available in different sizes and shapes. The most common types are cylindrical or conical. They are available in different diameters according to interdental space, ranging from 1.9 to 14mm. Selected brush should be slightly larger than the embrasure space. Introduction of brush in interdental space should be done obliquely, from the apical direction and used with back-and-forth motion. In type 2 embrasure patients, interdental brush is prescribed. It consists of soft nylon filaments twisted into a fine stainless steel wire. These interdental brushes are available in different sizes and shapes. The most common types are cylindrical or conical. They are available in different diameters according to interdental space, ranging from 1.9 to 14mm. Selected brush should be slightly larger than the embrasure space. Introduction of brush in interdental space should be done obliquely, from the apical direction and used with back-and-forth motion.

Use of mobile phone has increased globally; over half of world's 6.5 billion people use mobile phone services. wireless subscription in India stands at 952.34 million (in urban 553.45million whereas in rural 398.89) at the end of January 2015. Use of mobile technology to improve health outcomes is known as mobile health (mHealth). Text messages have become very common now and can be used to educate and motivate patients. Studies in medicine and dentistry have shown that text messaging is a very efficient tool for behavioral change and disease prevention. Use of mobile phone has increased globally; over half of world's 6.5 billion people use mobile phone services. wireless subscription in India stands at 952.34 million (in urban 553.45million whereas in rural 398.89) at the end of January 2015. Use of mobile technology to improve health outcomes is known as mobile health (mHealth). Text messages have become very common now and can be used to educate and motivate patients. Studies in medicine and dentistry have shown that text messaging is a very efficient tool for behavioral change and disease prevention.

The present prospective, randomized controlled clinical trial will be conducted in the department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences, Rohtak, Haryana. Duration of study will be 12 to 14 months and Patients will be recruited from the outpatient department of Periodontology. It will be divided into two groups, Test group will include scaling and root planing, interdental brushing demonstration and text messages in type 2 embrasure patients and Control group will include scaling and root planing, interdental brushing demonstration in type 2 embrasure patients.

All the participants will undergo phase 1 therapy with a combination of hand scalers and curettes and ultrasonic scaler. Standardized oral hygiene instructions will be imparted and will be reinforced at each appointment.

Most snugly fitted interdental brush will be selected and patient will be asked to pass interdental brush from buccal to lingual aspect of interdental area and then back out again while depressing the interdental papilla to allow bristles to reach sub-gingivally. Regular text messages twice a week, will be sent to the patients in the test group which will include reminder messages for interdental brushing. Patient will be asked to respond to messages.

Text message content for Reminder for using INTERDENTAL BRUSH

Primary outcome will include Plaque Index (Turesky modified Quigley & Hein) and Papillary Bleeding Index and secondary outcome will include Clinical attachment level (CAL), Gingival Index (GI), Pocket probing depth (PPD), Bleeding on probing (BOP), Interdental papilla height.

Papillary bleeding index will be measured at mesial and distal papilla of each tooth with Periodontal probe.

Plaque index will be measured on buccal and lingual surface with Periodontal probe.

Gingival index will be used to assess severity of gingival inflammation with the help of periodontal probe at 4 sites (Buccal, lingual, mesial and distal).

Clinical attachment level will be measured as the distance between the cemento-enamel junction and the base of pocket. Measurements will be made at 6 sites of each tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, and disto-lingual) using Periodontal probe.

Probing pocket depth will be measured as the distance from gingival margin to the base of pocket. Measurements will be noted at 6 sites of a tooth (mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual and disto-lingual).

Interdental papilla height will be measured as the distance from the tip of papilla to an imaginary line connecting most apical point of gingival zenith of adjacent teeth with the help of calibrated probe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 embrasures, with atleast 4 interdental spaces eligible for use of interdental brush.
* 2 or 3 periodontitis with probing pocket depth ≤5mm.
* Age - 30-55 years.
* Patients who own mobile phones.
* Patients who can read and write.
* No history of performing interdental oral hygiene on regular basis.
* Patients willing to comply with the given instructions regarding the use of interdental brush.

Exclusion Criteria:

* Smokers and orthodontic patients.
* Patient with systemic disease that can influence the outcome of therapy.
* Physically and mentally impaired patients.
* Patient on drugs associated with gingival overgrowth.
* Pregnant females.
* Patients on oral contraceptives or hormone replacement therapy.
* Overhanging restorations.
* Patients using any other cleaning aids like mouthwash.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Plaque Index | 6 months
  Quigley & Hein modification will be used which will measure the plaque level on buccal, labial and lingual surface of teeth with the help of disclosing agent.0 = no plaque
  1. = separate flecks of plaque at the cervical margin of the tooth
  2. = a thin continuous band of plaque (up to 1 mm) at the cervical margin
  3. = a band of plaque wider than 1 mm but covering less than 1/3 of crown
  4. = plaque covering at least 1 /3 but less than 2/3 of the crown
  5. = plaque covering 2/3 or more of crown
Papillary Bleeding Index | 6 months
  * Papillary bleeding index by Saxer et al will be used to assess gingival bleeding. A blunt periodontal probe was carefully inserted into the gingival sulcus at the base of the papilla on the mesial aspect, then moved coronally to the papilla tip. This was repeated on the distal aspect of the same papilla. The intensity of any bleeding thus provoked was recorded on a 0-4scale. Score 0 No bleeding Score 1- A single discreet bleeding point appears Score 2 - Several isolated bleeding points or a single fine line of blood appears
  Score 3 - The interdental triangle fills with blood shortly after probing Score 4- Profuse bleeding occurs after probing blood flows immediately into the marginal sulcus

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Yadav, BDS, Principal Investigator — Post graduate institute of dental sciences, Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yadav J, Tanwar N, Sharma RK, Sangwan A. Mobile Health to Improve Efficacy of Interdental Brushing Among Periodontitis Patients: A Randomized Clinical Trial. J Periodontal Res. 2025 Jun;60(6):559-569. doi: 10.1111/jre.13362. Epub 2024 Nov 25. PMID 39584464